CLINICAL TRIAL: NCT02382289
Title: Radiofrequency Ablation for the Treatment of Chronic Sacroiliac Joint Arthropathy; Comparing the Use of Bipolar RF at Six Points Versus Monopolar RF at Six Points and Three Points
Brief Title: Radiofrequency in Sacroiliac Arthropathy;Bipolar RF 6 Points Versus Monopolar RF at 6 and 3 Points
Acronym: RFSIBIMONO6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Hamad University Hospital, Bahrain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Mour2014/60
Record Dates: First submitted 2015-03-03; First posted 2015-03-06 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Radiofrequency Ablation; Chronic Sacroiliac Joint Arthropathy
Keywords: Radiofrequency; monopolar; bipolar; Sacroiliac Joint Arthropathy; three different modalities
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- bipolar RF 6 points (Active Comparator): Six RF needles will be put between the SIJ and the lateral aspects of the ipsilateral dorsal sacral foramina. After sensory and motor stimulation, bipolar lesion RF at 80oc for 90 sec will be applied between each successive pairs of needles.
  Interventions: Procedure: radiofrequency ablation for sacroiliac joint arthropathy
- monopolar RF 6 points (Active Comparator): RF needle is inserted at six levels in the area between the SIJ and the lateral aspects of the ipsilateral dorsal sacral foramina. after sensory and motor stimulation, monopolar lesion RF at 80oc for 90 sec will be applied.
  Interventions: Procedure: radiofrequency ablation for sacroiliac joint arthropathy
- monopolar RF 3 points (Active Comparator): RF needle is inserted at three levels in the upper , middle and lower part of the area between the SIJ and the lateral aspects of the ipsilateral dorsal sacral foramina. after sensory and motor stimulation, monopolar lesion RF at 80oc for 90 sec will be applied.
  Interventions: Procedure: radiofrequency ablation for sacroiliac joint arthropathy

INTERVENTIONS:
Procedure: radiofrequency ablation for sacroiliac joint arthropathy — comparing bipolar RF at 6 points with monopolar RF at 3 and 6 points for the treatment of SI arthropathy

SUMMARY:
Expecting using bipolar RF at six points, in spite of potentially consuming more intraoperative time, to be more effective and long lasting in the management of pain resultant from chronic sacroiliac joint arthropathy than the other 2 techniques using the monopolar RF even if using six points.

DETAILED DESCRIPTION:
A Prospective, single center, double blind, controlled randomized trial.

Sample Size:

Total of 60 patients divided into three groups:

Group 1: 20 patients will be receiving bipolar RF at six points. Group 2: 20 patients will be receiving monopolar RF at six points. Group 3: 20 patients will be receiving monopolar RF at three points.

Sampling technique:

Patients will be randomly divided in three groups. There will be a box with 60 closed envelopes, divided randomly in to three groups with 20 envelops in each group. On arrival to theatre one of the envelops will be opened and the assigned method will be applied.

Timeframe of the study:

6-12 months

Procedure:

After fulfilling inclusion criteria and apart from the exclusion criteria, patients will do either one of the three procedures according to the randomization. All patients will do the procedure under fluoroscopic guidance with use of Cosman RF generator G4TM, 20 gauge straight sharp cannula, 10 cm shaft, 10 mm tip and 10 cm electrodes (Cosman autoclavable CSK-TC10).

Group 1 ; Six RF needles will be put between the SIJ and the lateral aspects of the ipsilateral dorsal sacral foramina. After sensory and motor stimulation, bipolar lesion RF at 80oc for 90 sec will be applied between each successive pairs of needles.

Group 2; RF needle is inserted at six levels in the area between the SIJ and the lateral aspects of the ipsilateral dorsal sacral foramina. after sensory and motor stimulation, monopolar lesion RF at 80oc for 90 sec will be applied.

Group 3; RF needle is inserted at six levels in the upper , middle and lower part of the area between the SIJ and the lateral aspects of the ipsilateral dorsal sacral foramina. after sensory and motor stimulation, monopolar lesion RF at 80oc for 90 sec will be applied.

Patients will be evaluated by a specialized pain nurse after 2 weeks, one month, 3 months and 6 months for pain score using the visual analogue pain scale.

Overall patient satisfaction with pain relief will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* • Moderate to severe low back pain for more than six months with positive Patrick's and Yeoman's tests with tenderness over the SI joint.

  * Pain is not responding to the usual medical treatment.
  * More than 50 % pain relief after diagnostic injection with local anesthetic.

Exclusion Criteria:

* • Patient refusal to do the procedure or to share in the study

  * Focal Neurologic Signs.
  * significant anticoagulation e.g. clopedogril (low dose aspirin will be excluded)
  * Pregnancy, breast feeding or planning on becoming pregnant during the trial.
  * Infection at the intended injection site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
patient satisfaction | 6-12 months
  Patients suffering chronic low back pain due to sacroiliac joint arthropathy will receive a potentially more effective method of radiofrequency ablation with an overall better patient satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: mohamed hashim, SR anesthesia, Principal Investigator
Locations (1):
- King Hamad University Hospital, Muharraq, Manama, Bahrain